CLINICAL TRIAL: NCT02323295
Title: Pilot Study of the Effect of High Doses of Radiation on Bone Metabolism and Structure in Patients Treated With Adjuvant Radiotherapy and Surgery for Sacral Tumors
Brief Title: Effect of High Doses of Radiation on Bone Structure and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Schwab, Joseph H., Instructor in Orthopaedic Surgery, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-208; C06CA059267 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-12-23 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Malignant Bone Tumors
Keywords: Malignant bone tumors
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non Surgical-Radiation Only (Experimental): Non-surgical candidates receive 72 up to 77.l4 Gy of radiation depending on the histology (72 Gy for osteosarcoma and chondrosarcoma and 77.4 Gy for chordoma
  Interventions: Radiation: Radiation (Non-surgical Arm)
- Malignant Tumor Surgery And Radiation (Experimental): The standard treatment includes pre-operative radiation of 50.4 Gy, followed by a recovery period of approximately 4 to 5 weeks. Surgery involves removing the malignant tumor in the sacrum in one piece, preferably with a cuff of normal tissue around the tumor. After approximately 6 weeks of recovery, the patient is treated with another 19.8 Gy up to 27 Gy of radiation postoperatively depending on the final margin status (higher for gross residual disease). If the wound is not healed or there is another medical reason to delay adjuvant radiation, then radiation may begin later.
  Interventions: Radiation: Radiation (Surgical Arm); Procedure: Malignant Tumor Surgery

INTERVENTIONS:
Radiation: Radiation (Surgical Arm) — For surgical candidates, the standard treatment includes pre-operative radiation of 50.4 Gy, followed by a recovery period of approximately 4 to 5 weeks. After this surgery will take place. After approximately 6 weeks of recovery, to allow the surgical incision to heal, the patient is treated with another 19.8 Gy up to 27 Gy of radiation postoperatively depending on the final margin status (higher for gross residual disease)
  Arms: Malignant Tumor Surgery And Radiation
Radiation: Radiation (Non-surgical Arm) — Non-surgical candidates receive 72 up to 77.14 Gy of radiation depending on the histology (72 Gy for osteosarcoma and chondrosarcoma and 77.4 Gy for chordoma)
  Arms: Non Surgical-Radiation Only
Procedure: Malignant Tumor Surgery — Surgery involves removing the malignant tumor in the sacrum in one piece, preferably with a cuff of normal tissue around the tumor
  Arms: Malignant Tumor Surgery And Radiation

SUMMARY:
This study is designed to characterize the effects of high energy radiation on bone breakdown, with a specific interest in reducing the rate of sacral fractures. Although radiation is very important in managing tumors, it is related to complications such as bone fractures. In this research study, the investigators are looking to determine changes in blood markers, bone density, and bone structure following radiation and to better understand the reason for these changes.

DETAILED DESCRIPTION:
Participants in the Surgical Arm of the study will be treated according to the schedule outlined in protocol for a combined treatment with surgery and adjuvant high dose radiotherapy. Patients in the non surgical arm of the the study will be treated according to the protocol being treated with radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* All laboratory tests that are a part of the eligibility criteria must be completed within 14 days prior to the date of registration. Diagnostic tests that are a part of the eligibility criteria must be performed within 30 days of the date of registration. Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Study participants must have histologically confirmed primary malignant bone tumor in the sacrum for which surgery and radiation or radiation alone are planned.
* Age 18 years or older. In children under the age of 8, tetracycline derivatives have been reported to stain tooth enamel yellow color. These considerations lead us to exclude young persons under the age of 18 from the study.
* Participants must have normal organ and marrow function as defined below:

  * Total bilirubin within normal institutional limits
  * Aspartaataminotransferase (AST) (SGOT)/ Alanine-aminotransferase (ALT) (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal limit
* The effects of tetracyclines and radiation used in computer tomography on the developing human fetus are known to be detrimental. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Participants must be able to read and understand English language and have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Participants who have had surgery, chemotherapy, or radiotherapy of the sacrum prior to entering the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tetracyclines.
* Pregnant or nursing
* Uncontrolled inter current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Schwab, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Surgical-Radiation Only: Non-surgical candidates receive 72 up to 77.l4 Gy of radiation depending on the histology (72 Gy for osteosarcoma and chondrosarcoma and 77.4 Gy for chordoma
  Radiation: For surgical candidates, the standard treatment includes pre-operative radiation of 50.4 Gy, followed by a recovery period of approximately 4 to 5 weeks. After this surgery will take place. After approximately 6 weeks of recovery, to allow the surgical incision to heal, the patient is treated with another 19.8 Gy up to 27 Gy of radiation postoperatively depending on the final margin status (higher for gross residual disease) Non-surgical candidates receive 72 up to 77.14 Gy of radiation depending on the histology (72 Gy for osteosarcoma and chondrosarcoma and 77.4 Gy for chordoma)
- Malignant Tumor Surgery And Radiation: The standard treatment includes pre-operative radiation of 50.4 Gy, followed by a recovery period of approximately 4 to 5 weeks. Surgery involves removing the malignant tumor in the sacrum in one piece, preferably with a cuff of normal tissue around the tumor. After approximately 6 weeks of recovery, the patient is treated with another 19.8 Gy up to 27 Gy of radiation postoperatively depending on the final margin status (higher for gross residual disease). If the wound is not healed or there is another medical reason to delay adjuvant radiation, then radiation may begin later.
  Radiation: For surgical candidates, the standard treatment includes pre-operative radiation of 50.4 Gy, followed by a recovery period of approximately 4 to 5 weeks. After this surgery will take place. After approximately 6 weeks of recovery, to allow the surgical incision to heal, the patient is treated with another 19.8 Gy up to 27 Gy of radiation postoperatively depending on the final margin status (higher for gross residual disease) Non-surgical candidates receive 72 up to 77.14 Gy of radiation depending on the histology (72 Gy for osteosarcoma and chondrosarcoma and 77.4 Gy for chordoma)
  Malignant Tumor Surgery: Surgery involves removing the malignant tumor in the sacrum in one piece, preferably with a cuff of normal tissue around the tumor
Period: Overall Study
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Started | 2 | 10
Completed | 2 | 7
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Patient did not have surgery as planned. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation | Total
Number analyzed (Participants) | 2 | 10 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 9 | 10
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 10 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 10 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (Tb. BMD)
Description: Trabecular bone mineral density will be measured in mg/cm3 using volumetric Quantitative Computed Tomography (QCT) of L1, L2 and the vertebrae adjacent to the tumor.
Time Frame: Non-surgical arm: baseline, 3 months Surgical arm: baseline, 9 weeks
Population: Subjects 4 and 9 are in the non-surgical radiation group and only have values for that column. The rest of the subjects are in the malignant tumor surgery and radiation and only have values in that column.
Measure: Number; unit: mg/cm^3
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
mg/cm^3
  Subject 2 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 2 (lumbar) |  | 4.5
  Subject 2 (sacral): number analyzed (Participants) | 0 | 1
  Subject 2 (sacral) |  | -39.3
  Subject 3 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 3 (lumbar) |  | -8.7
  Subject 3 (sacral): number analyzed (Participants) | 0 | 1
  Subject 3 (sacral) |  | -54.7
  Subject 4 (lumbar): number analyzed (Participants) | 1 | 0
  Subject 4 (lumbar) | 4.1 |
  Subject 4 (sacral): number analyzed (Participants) | 1 | 0
  Subject 4 (sacral) | 5.2 |
  Subject 6 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 6 (lumbar) |  | -2.6
  Subject 6 (sacral): number analyzed (Participants) | 0 | 1
  Subject 6 (sacral) |  | -32.7
  Subject 7 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 7 (lumbar) |  | 3.6
  Subject 7 (sacral): number analyzed (Participants) | 0 | 1
  Subject 7 (sacral) |  | -14.8
  Subject 8 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 8 (lumbar) |  | -2.2
  Subject 8 (sacral): number analyzed (Participants) | 0 | 1
  Subject 8 (sacral) |  | -57.7
  Subject 9 (lumbar): number analyzed (Participants) | 1 | 0
  Subject 9 (lumbar) | -3.5 |
  Subject 9 (sacral): number analyzed (Participants) | 1 | 0
  Subject 9 (sacral) | -55.7 |
  Subject 10 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 10 (lumbar) |  | -0.2
  Subject 10 (sacral): number analyzed (Participants) | 0 | 1
  Subject 10 (sacral) |  | -70.3
  Subject 12 (lumbar): number analyzed (Participants) | 0 | 1
  Subject 12 (lumbar) |  | 3.3
  Subject 12 (sacral): number analyzed (Participants) | 0 | 1
  Subject 12 (sacral) |  | -37.9

2. Secondary Outcome: Serum N-Telopeptide (NTX)
Description: Indicator for Bone Formation, units reported in nmol NTX/mmol creatinine
Time Frame: Non-surgical arm: baseline, 3.5 weeks, 7 weeks, ~5 months, ~8 months Surgical arm: baseline, 5.5 weeks, 18.5 weeks, ~7 months, ~10 months
Population: Subjects 4 and 9 are in the non-surgical radiation group and only have values for that column. The rest of the subjects are in the malignant tumor surgery and radiation and only have values in that column.
  For other missing values, certain tests were not performed at certain timepoints for some subjects.
Measure: Number; unit: nM/L
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
nM/L
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 21.711
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 17.76
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 31.447
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 24.376
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 21.889
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 11.217
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 14.294
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 4.614 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 7.366 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 6.205 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 7.218 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 15.932
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 19.973
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 20.922
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 16.707
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 14.096
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 15.949
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 8.942
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 25.817
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 18.513
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 11.97
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 19.065
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 22.917
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 26.767
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 18.116
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 8.028 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 12.435 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 7.642 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 11.163 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 11.155 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 11.082
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 7.763
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 10.123
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 9.89
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 12.656
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 10.511
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 14.693
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 15.177
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Serum Tartrate-resistant Acid Phosphatase 5b (TRAP5b)
Description: Indicator for Bone Formation, units reported in U/L
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: U/L
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
U/L
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 3.823813
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 3.503794
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 4.465143
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 4.226845
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 3.87936
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 4.235948
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 5.111555
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 2.951546 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 3.597596 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 3.22168 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 2.830882 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 5.482747
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 4.700929
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 6.675976
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 4.910525
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 3.99912
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 5.051881
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 4.211249
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 5.499551
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 3.725495
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 3.890646
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 4.353515
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 5.2026
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 5.025804
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 3.984603
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 2.461792 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 2.601314 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 3.056594 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 3.203289 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 2.194518 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 3.122802
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 2.776157
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 3.329006
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 2.496301
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 3.702653
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 3.986177
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 3.969791
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 3.615732
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serum Osteocalcin (OC)
Description: Indicator for Bone Formation, units reported in ng/mL
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: ng/mL
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
ng/mL
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 14.304331
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 14.398441
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 39.41674
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 24.231676
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 18.05678
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 31.395938
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 16.128416
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 7.70232 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 8.504592 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 10.025644 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 10.54423 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 10.954567
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 12.869497
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 13.061037
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 25.763047
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 18.419998
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 4.378182
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 10.369156
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 40.882969
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 28.262384
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 13.966
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 16.786965
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 32.353007
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 29.73705
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 26.099775
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 12.220099 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 12.368649 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 10.955072 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 11.167479 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 10.028165 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 12.321595
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 14.881427
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 19.861684
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 16.437832
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 17.549564
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 17.154958
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 11.480525
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 16.409198
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serum Type 1 Procollagen N-terminal (P1NP)
Description: Indicator for systemic metabolism that can affect bone health, units reported in pg/mL
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: pg/mL
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
pg/mL
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 42.826123
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 34.128407
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 123.860111
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 74.655436
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 68.966468
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 72.946381
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 44.08789
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 21.375865 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 28.095207 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 32.953174 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 43.37268 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 129.054174
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 83.031563
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 152.713648
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 186.103683
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 93.061044
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 13.875913
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 40.4564
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 135.28581
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 98.31769
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 39.183829
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 56.609907
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 219.86073
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 129.372101
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 99.637646
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 51.29302 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 38.642487 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 40.145122 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 42.945924 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 33.200638 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 53.568154
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 59.57128
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 114.083432
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 59.498204
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 47.539351
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 50.82762
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 72.878306
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 64.002627
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Serum Phosphate (P)
Description: Indicators for systemic metabolism that can affect bone health, units reported in mg/dL
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mg/dL
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
mg/dL
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 3.9
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 3.5
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 4.0
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 3.6
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 3.7
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 4.4
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 4.3
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 2.8 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 3.0 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 3.0 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 3.2 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 3.4
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 3.3
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 4.4
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 4.1
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 3.6
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 3.3
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 4.0
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 4.9
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 4.0
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 3.3
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 3.3
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 3.5
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 3.7
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 3.3
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 4.3 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 4.0 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 4.7 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 4.2 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 3.4 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 2.4
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 4.0
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 3.5
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 2.2
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 4.2
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 3.7
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 3.4
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 3.4
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serum 25-hydroxycalciferol Vit D (25-OH VitD)
Description: Indicators for systemic metabolism that can affect bone health, units reported in nmol/L
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: nmol/L
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 2 | 7
nmol/L
  Subject 2 (baseline): number analyzed (Participants) | 0 | 1
  Subject 2 (baseline) |  | 36.065991
  Subject 2 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (5.5 weeks) |  | 32.073769
  Subject 2 (18.5 Weeks): number analyzed (Participants) | 0 | 1
  Subject 2 (18.5 Weeks) |  | 31.302671
  Subject 2 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 7 months) |  | 36.77789
  Subject 2 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 2 (about 10 months) |  | 33.419347
  Subject 3 (baseline): number analyzed (Participants) | 0 | 1
  Subject 3 (baseline) |  | 17.038722
  Subject 3 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 3 (5.5 weeks) |  | 12.739664
  Subject 3 (18.5 weeks): number analyzed (Participants) | 0 | 0
  Subject 3 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 3 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 4 (baseline): number analyzed (Participants) | 1 | 0
  Subject 4 (baseline) | 60.483526 |
  Subject 4 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (3.5 weeks) | 50.942045 |
  Subject 4 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 4 (7 weeks) | 38.703589 |
  Subject 4 (about 5 months): number analyzed (Participants) | 0 | 0
  Subject 4 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 4 (about 8 months) | 62.317379 |
  Subject 6 (baseline): number analyzed (Participants) | 0 | 1
  Subject 6 (baseline) |  | 36.051246
  Subject 6 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (5.5 weeks) |  | 35.309918
  Subject 6 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 6 (18.5 weeks) |  | 36.748899
  Subject 6 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 7 months) |  | 32.918895
  Subject 6 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 6 (about 10 months) |  | 36.262804
  Subject 7 (baseline): number analyzed (Participants) | 0 | 1
  Subject 7 (baseline) |  | 17.740625
  Subject 7 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (5.5 weeks) |  | 17.258697
  Subject 7 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 7 (18.5 weeks) |  | 27.862934
  Subject 7 (about 7 months): number analyzed (Participants) | 0 | 0
  Subject 7 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 7 (about 10 months) |  | 20.845497
  Subject 8 (baseline): number analyzed (Participants) | 0 | 1
  Subject 8 (baseline) |  | 23.596514
  Subject 8 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (5.5 weeks) |  | 22.190329
  Subject 8 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 8 (18.5 weeks) |  | 27.355142
  Subject 8 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 7 months) |  | 29.649107
  Subject 8 (about 10 months): number analyzed (Participants) | 0 | 1
  Subject 8 (about 10 months) |  | 25.399281
  Subject 9 (baseline): number analyzed (Participants) | 1 | 0
  Subject 9 (baseline) | 39.515148 |
  Subject 9 (3.5 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (3.5 weeks) | 39.281166 |
  Subject 9 (7 weeks): number analyzed (Participants) | 1 | 0
  Subject 9 (7 weeks) | 40.21479 |
  Subject 9 (about 5 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 5 months) | 41.193903 |
  Subject 9 (about 8 months): number analyzed (Participants) | 1 | 0
  Subject 9 (about 8 months) | 47.316427 |
  Subject 10 (baseline): number analyzed (Participants) | 0 | 1
  Subject 10 (baseline) |  | 30.093394
  Subject 10 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (5.5 weeks) |  | 30.491835
  Subject 10 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 10 (18.5 weeks) |  | 27.330808
  Subject 10 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 10 (about 7 months) |  | 28.958284
  Subject 10 (about 10 months): number analyzed (Participants) | 0 | 0
  Subject 12 (baseline): number analyzed (Participants) | 0 | 1
  Subject 12 (baseline) |  | 18.366566
  Subject 12 (5.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (5.5 weeks) |  | 25.333837
  Subject 12 (18.5 weeks): number analyzed (Participants) | 0 | 1
  Subject 12 (18.5 weeks) |  | 31.425202
  Subject 12 (about 7 months): number analyzed (Participants) | 0 | 1
  Subject 12 (about 7 months) |  | 32.557435
  Subject 12 (about 10 months): number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mineral Apposition Rate (MAR)
Description: Tetracycline quadruple labeling method will be used and the unit of measure will be um/day
Time Frame: Only surgical arm: The months after biopsies are taken during surgery (surgery is during week 4 and 5). These measurements will be done in batches so timeframe isn't clear.
Population: B = before radiation, A = after radiation. For missing values, certain tests were not performed at certain timepoints for some subjects.
Measure: Number; unit: um/day
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
um/day
  Subject 2 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Cancellous, B) |  | 0.64
  Subject 2 (iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (iliac Crest, Cancellous, A) |  | 0.66
  Subject 2 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Endocortical, B) |  | 0.55
  Subject 2 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Endocortical, A) |  | 0.71
  Subject 2 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Intracortical, B) |  | 0.72
  Subject 2 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Intracortical, A) |  | 0.44
  Subject 2 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 2 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 2 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Cancellous, B) |  | 0.58
  Subject 2 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Cancellous, A) |  | 0.45
  Subject 2 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Endocortical, B) |  | 0.70
  Subject 2 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 2 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Intracortical, B) |  | 0.47
  Subject 2 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 2 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Periosteal, B) |  | 1.50
  Subject 2 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Periosteal, A) |  | 0.98
  Subject 3 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Cancellous, B) |  | 0.64
  Subject 3 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Cancellous, A) |  | 0.54
  Subject 3 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Endocortical, B) |  | 0.53
  Subject 3 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Endocortical, A) |  | 0.46
  Subject 3 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Intracortical, B) |  | 0.64
  Subject 3 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Intracortical, A) |  | 0.59
  Subject 3 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Sacrum, Cancellous, B) |  | 0.62
  Subject 3 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Sacrum, Cancellous, A) |  | 0.34
  Subject 3 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 6 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Cancellous, B) |  | 0.51
  Subject 6 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Cancellous, A) |  | 0.40
  Subject 6 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Endocortical, B) |  | 0.51
  Subject 6 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Endocortical, A) |  | 0.43
  Subject 6 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Intracortical, B) |  | 1.12
  Subject 6 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Intracortical, A) |  | 0.50
  Subject 6 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 6 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 6 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Cancellous, B) |  | 0.51
  Subject 6 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Cancellous, A) |  | 0.37
  Subject 6 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Endocortical, B) |  | 0.55
  Subject 6 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Endocortical, A) |  | 0.18
  Subject 6 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 0
  Subject 6 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 6 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 6 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Cancellous, B) |  | 0.65
  Subject 7 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Cancellous, A) |  | 0.72
  Subject 7 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Endocortical, A) |  | 0.48
  Subject 7 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Intracortical, B) |  | 1.20
  Subject 7 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Periosteal, B) |  | 0.33
  Subject 7 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Periosteal, A) |  | 0.47
  Subject 7 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Cancellous, B) |  | 0.69
  Subject 7 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Cancellous, A) |  | 0.59
  Subject 7 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Endocortical, B) |  | 0.41
  Subject 7 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Endocortical, A) |  | 0.76
  Subject 7 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Intracortical, B) |  | 0.92
  Subject 7 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Intracortical, A) |  | 0.68
  Subject 7 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 7 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Cancellous, B) |  | 0.62
  Subject 8 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Cancellous, A) |  | 0.43
  Subject 8 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Endocortical, B) |  | 0.51
  Subject 8 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Endocortical, A) |  | 0.33
  Subject 8 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Intracortical, B) |  | 1.83
  Subject 8 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Intracortical, A) |  | 0.73
  Subject 8 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Sacrum, Cancellous, B) |  | 0.56
  Subject 8 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Cancellous, B) |  | 0.60
  Subject 10 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Cancellous, A) |  | 0.40
  Subject 10 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Endocortical, B) |  | 0.42
  Subject 10 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Endocortical, A) |  | 0.41
  Subject 10 (Iliac Crest, Intracortical, B) |  | 0.49
  Subject 10 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Intracortical, A) |  | 0.53
  Subject 10 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 10 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Cancellous, B) |  | 0.50
  Subject 10 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Cancellous, A) |  | 0.49
  Subject 10 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Endocortical, B) |  | 0.44
  Subject 10 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Intracortical, B) |  | 0.60
  Subject 10 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Cancellous, B) |  | 0.53
  Subject 12 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Endocortical, B) |  | 0.48
  Subject 12 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Intracortical, B) |  | 0.96
  Subject 12 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Cancellous, B) |  | 0.47
  Subject 12 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Endocortical, B) |  | 0.50
  Subject 12 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Intracortical, B) |  | 1.31
  Subject 12 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Bone Formation Rate (BFR/BS)
Description: Tetracycline quadruple labeling method will be used and the unit of measure will be mm3/mm2/year
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number; unit: mm3/mm2/year
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
mm3/mm2/year
  Subject 2 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Cancellous, B) |  | 0.003
  Subject 2 (iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (iliac Crest, Cancellous, A) |  | 0.003
  Subject 2 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Endocortical, B) |  | 0.013
  Subject 2 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Endocortical, A) |  | 0.013
  Subject 2 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Intracortical, B) |  | 0.014
  Subject 2 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Intracortical, A) |  | 0.013
  Subject 2 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Periosteal, B) |  | 0.000
  Subject 2 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Periosteal, A) |  | 0.000
  Subject 2 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Cancellous, B) |  | 0.007
  Subject 2 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Cancellous, A) |  | 0.001
  Subject 2 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Endocortical, B) |  | 0.052
  Subject 2 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 2 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Intracortical, B) |  | 0.053
  Subject 2 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Intracortical, A) |  | 0.000
  Subject 2 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Periosteal, B) |  | 0.012
  Subject 2 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Periosteal, A) |  | 0.004
  Subject 3 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Cancellous, B) |  | 0.016
  Subject 3 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Cancellous, A) |  | 0.012
  Subject 3 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Endocortical, B) |  | 0.021
  Subject 3 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Endocortical, A) |  | 0.009
  Subject 3 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Intracortical, B) |  | 0.047
  Subject 3 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Intracortical, A) |  | 0.032
  Subject 3 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Periosteal, B) |  | 0.000
  Subject 3 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Periosteal, A) |  | 0.000
  Subject 3 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 3 (Sacrum, Cancellous, B) |  | 0.009
  Subject 3 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Sacrum, Cancellous, A) |  | 0.001
  Subject 3 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 6 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Cancellous, B) |  | 0.005
  Subject 6 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Cancellous, A) |  | 0.006
  Subject 6 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Endocortical, B) |  | 0.019
  Subject 6 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Endocortical, A) |  | 0.024
  Subject 6 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Intracortical, B) |  | 0.029
  Subject 6 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Intracortical, A) |  | 0.041
  Subject 6 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Periosteal, B) |  | 0.000
  Subject 6 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Periosteal, A) |  | 0.000
  Subject 6 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Cancellous, B) |  | 0.003
  Subject 6 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Cancellous, A) |  | 0.001
  Subject 6 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Endocortical, B) |  | 0.010
  Subject 6 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Endocortical, A) |  | 0.001
  Subject 6 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Intracortical, B) |  | 0.000
  Subject 6 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Intracortical, A) |  | 0.000
  Subject 6 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Periosteal, B) |  | 0.000
  Subject 6 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Periosteal, A) |  | 0.000
  Subject 7 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Cancellous, B) |  | 0.012
  Subject 7 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Cancellous, A) |  | 0.031
  Subject 7 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Endocortical, A) |  | 0.004
  Subject 7 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Intracortical, B) |  | 0.057
  Subject 7 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Periosteal, B) |  | 0.007
  Subject 7 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Periosteal, A) |  | 0.036
  Subject 7 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Cancellous, B) |  | 0.011
  Subject 7 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Cancellous, A) |  | 0.007
  Subject 7 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Endocortical, B) |  | 0.004
  Subject 7 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Endocortical, A) |  | 0.007
  Subject 7 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Intracortical, B) |  | 0.004
  Subject 7 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Intracortical, A) |  | 0.002
  Subject 7 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Periosteal, B) |  | 0.000
  Subject 7 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Periosteal, A) |  | 0.000
  Subject 8 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Cancellous, B) |  | 0.004
  Subject 8 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Cancellous, A) |  | 0.001
  Subject 8 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Endocortical, B) |  | 0.016
  Subject 8 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Endocortical, A) |  | 0.007
  Subject 8 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Intracortical, B) |  | 0.039
  Subject 8 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Intracortical, A) |  | 0.035
  Subject 8 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Periosteal, B) |  | 0.000
  Subject 8 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Periosteal, A) |  | 0.000
  Subject 8 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 8 (Sacrum, Cancellous, B) |  | 0.005
  Subject 8 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Cancellous, B) |  | 0.022
  Subject 10 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Cancellous, A) |  | 0.016
  Subject 10 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Endocortical, B) |  | 0.022
  Subject 10 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Endocortical, A) |  | 0.030
  Subject 10 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Intracortical, B) |  | 0.023
  Subject 10 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Intracortical, A) |  | 0.032
  Subject 10 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Periosteal, B) |  | 0.000
  Subject 10 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Periosteal, A) |  | 0.000
  Subject 10 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Cancellous, B) |  | 0.003
  Subject 10 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Cancellous, A) |  | 0.001
  Subject 10 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Endocortical, B) |  | 0.002
  Subject 10 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Intracortical, B) |  | 0.013
  Subject 10 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Periosteal, B) |  | 0.000
  Subject 10 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Periosteal, A) |  | 0.000
  Subject 12 (Iliac Crest, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Cancellous, B) |  | 0.018
  Subject 12 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Endocortical, B) |  | 0.028
  Subject 12 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Iliac Crest, Intracortical, B) |  | 0.017
  Subject 12 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Periosteal, B): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Periosteal, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Cancellous, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Cancellous, B) |  | 0.005
  Subject 12 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Endocortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Endocortical, B) |  | 0.017
  Subject 12 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Intracortical, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Intracortical, B) |  | 0.063
  Subject 12 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Periosteal, B): number analyzed (Participants) | 0 | 1
  Subject 12 (Sacrum, Periosteal, B) |  | 0.000
  Subject 12 (Sacrum, Periosteal, A): number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mineralization Lag Time (Mlt)
Description: Tetracycline quadruple labeling method will be used and the unit of measure will be days
Time Frame: as for outcome 8
Population: A = after radiation. No periosteal data for any subject. For other missing values, certain tests were not performed at certain timepoints for some subjects.
Measure: Number; unit: days
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
days
  Subject 2 (iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (iliac Crest, Cancellous, A) |  | 40.77
  Subject 2 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Endocortical, A) |  | 15.47
  Subject 2 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Iliac Crest, Intracortical, A) |  | 12.56
  Subject 2 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 2 (Sacrum, Cancellous, A) |  | 68.10
  Subject 2 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 2 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Cancellous, A) |  | 21.70
  Subject 3 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Endocortical, A) |  | 41.88
  Subject 3 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Iliac Crest, Intracortical, A) |  | 20.33
  Subject 3 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 3 (Sacrum, Cancellous, A) |  | 7.45
  Subject 3 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 3 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 6 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Cancellous, A) |  | 24.98
  Subject 6 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Endocortical, A) |  | 13.31
  Subject 6 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Iliac Crest, Intracortical, A) |  | 16.36
  Subject 6 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Cancellous, A) |  | 110.51
  Subject 6 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 6 (Sacrum, Endocortical, A) |  | 40.28
  Subject 6 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 7 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Cancellous, A) |  | 16.28
  Subject 7 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Iliac Crest, Endocortical, A) |  | 15.49
  Subject 7 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 7 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Cancellous, A) |  | 34.10
  Subject 7 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Endocortical, A) |  | 37.18
  Subject 7 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 7 (Sacrum, Intracortical, A) |  | 87.15
  Subject 8 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Cancellous, A) |  | 3.11
  Subject 8 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Endocortical, A) |  | 10.72
  Subject 8 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 8 (Iliac Crest, Intracortical, A) |  | 8.15
  Subject 8 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 8 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Cancellous, A) |  | 63.18
  Subject 10 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Endocortical, A) |  | 34.23
  Subject 10 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Iliac Crest, Intracortical, A) |  | 26.65
  Subject 10 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 1
  Subject 10 (Sacrum, Cancellous, A) |  | 142.08
  Subject 10 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 10 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Iliac Crest, Intracortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Cancellous, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Endocortical, A): number analyzed (Participants) | 0 | 0
  Subject 12 (Sacrum, Intracortical, A): number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Osteoblast Number (N.Ob/BPm)
Description: Immunohistochemistry staining methods will be used and the unit of measure will be mm^-1
Time Frame: Only surgical arm: The weeks after biopsies are taken during surgery (surgery is during week 4 and 5).
Population: No biopsy data for subjects 10 and 12.
Measure: Number; unit: 1/mm
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
1/mm
  Subject 2 (week 5): number analyzed (Participants) | 0 | 1
  Subject 2 (week 5) |  | 0.26
  Subject 2 (week 6): number analyzed (Participants) | 0 | 1
  Subject 2 (week 6) |  | 0.05
  Subject 3 (week 5): number analyzed (Participants) | 0 | 1
  Subject 3 (week 5) |  | 1.25
  Subject 3 (week 6): number analyzed (Participants) | 0 | 1
  Subject 3 (week 6) |  | 0.05
  Subject 6 (week 5): number analyzed (Participants) | 0 | 1
  Subject 6 (week 5) |  | 1.04
  Subject 6 (week 6): number analyzed (Participants) | 0 | 1
  Subject 6 (week 6) |  | 0.19
  Subject 7 (week 5): number analyzed (Participants) | 0 | 1
  Subject 7 (week 5) |  | 6.23
  Subject 7 (week 6): number analyzed (Participants) | 0 | 1
  Subject 7 (week 6) |  | 1.89
  Subject 8 (week 5): number analyzed (Participants) | 0 | 1
  Subject 8 (week 5) |  | 0.05
  Subject 8 (week 6): number analyzed (Participants) | 0 | 1
  Subject 8 (week 6) |  | 0.16
  Subject 10 (week 5): number analyzed (Participants) | 0 | 0
  Subject 10 (week 6): number analyzed (Participants) | 0 | 0
  Subject 12 (week 5): number analyzed (Participants) | 0 | 0
  Subject 12 (week 6): number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Osteoblast Surface (Ob. S/BS)
Description: Immunohistochemistry staining methods will be used and the unit of measure will be mm^-1
Time Frame: Only surgical arm: The weeks after biopsies are taken during surgery (surgery is during week 4 and 5).
Population: No biopsy data for subjects 10 and 12.
Measure: Number; unit: 1/mm
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
1/mm
  Subject 2 (week 5): number analyzed (Participants) | 0 | 1
  Subject 2 (week 5) |  | 0.58
  Subject 2 (week 6): number analyzed (Participants) | 0 | 1
  Subject 2 (week 6) |  | 0.10
  Subject 3 (week 5): number analyzed (Participants) | 0 | 1
  Subject 3 (week 5) |  | 2.38
  Subject 3 (week 6): number analyzed (Participants) | 0 | 1
  Subject 3 (week 6) |  | 0.07
  Subject 6 (week 5): number analyzed (Participants) | 0 | 1
  Subject 6 (week 5) |  | 1.63
  Subject 6 (week 6): number analyzed (Participants) | 0 | 1
  Subject 6 (week 6) |  | 0.29
  Subject 7 (week 5): number analyzed (Participants) | 0 | 1
  Subject 7 (week 5) |  | 9.07
  Subject 7 (week 6): number analyzed (Participants) | 0 | 1
  Subject 7 (week 6) |  | 2.71
  Subject 8 (week 5): number analyzed (Participants) | 0 | 1
  Subject 8 (week 5) |  | 0.05
  Subject 8 (week 6): number analyzed (Participants) | 0 | 1
  Subject 8 (week 6) |  | 0.23
  Subject 10 (week 5): number analyzed (Participants) | 0 | 0
  Subject 10 (week 6): number analyzed (Participants) | 0 | 0
  Subject 12 (week 5): number analyzed (Participants) | 0 | 0
  Subject 12 (week 6): number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Osteoclast Number (N.Oc/BPm)
Description: Immunohistochemistry staining methods will be used and the unit of measure will be mm^-1
Time Frame: Only surgical arm: The weeks after biopsies are taken during surgery (surgery is during week 4 and 5).
Population: No biopsy data for subjects 10 and 12.
Measure: Number; unit: 1/mm
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
1/mm
  Subject 2 (week 5): number analyzed (Participants) | 0 | 1
  Subject 2 (week 5) |  | 0.02
  Subject 2 (week 6): number analyzed (Participants) | 0 | 1
  Subject 2 (week 6) |  | 0.00
  Subject 3 (week 5): number analyzed (Participants) | 0 | 1
  Subject 3 (week 5) |  | 0.03
  Subject 3 (week 6): number analyzed (Participants) | 0 | 1
  Subject 3 (week 6) |  | 0.01
  Subject 6 (week 5): number analyzed (Participants) | 0 | 1
  Subject 6 (week 5) |  | 0.08
  Subject 6 (week 6): number analyzed (Participants) | 0 | 1
  Subject 6 (week 6) |  | 0.02
  Subject 7 (week 5): number analyzed (Participants) | 0 | 1
  Subject 7 (week 5) |  | 0.10
  Subject 7 (week 6): number analyzed (Participants) | 0 | 1
  Subject 7 (week 6) |  | 0.31
  Subject 8 (week 5): number analyzed (Participants) | 0 | 1
  Subject 8 (week 5) |  | 0
  Subject 8 (week 6): number analyzed (Participants) | 0 | 1
  Subject 8 (week 6) |  | 0.07
  Subject 10 (week 5): number analyzed (Participants) | 0 | 0
  Subject 10 (week 6): number analyzed (Participants) | 0 | 0
  Subject 12 (week 5): number analyzed (Participants) | 0 | 0
  Subject 12 (week 6): number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Osteoclast Surface (Oc.S/BS)
Description: Immunohistochemistry staining methods will be used and the unit of measure will be mm^-1
Time Frame: Only surgical arm: The weeks after biopsies are taken during surgery (surgery is during week 4 and 5).
Population: No biopsy data for subjects 10 and 12.
Measure: Number; unit: 1/mm
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
Number analyzed (Participants) | 0 | 7
1/mm
  Subject 2 (week 5): number analyzed (Participants) | 0 | 1
  Subject 2 (week 5) |  | 0.12
  Subject 2 (week 6): number analyzed (Participants) | 0 | 1
  Subject 2 (week 6) |  | 0.00
  Subject 3 (week 5): number analyzed (Participants) | 0 | 1
  Subject 3 (week 5) |  | 0.11
  Subject 3 (week 6): number analyzed (Participants) | 0 | 1
  Subject 3 (week 6) |  | 0.02
  Subject 6 (week 5): number analyzed (Participants) | 0 | 1
  Subject 6 (week 5) |  | 0.36
  Subject 6 (week 6): number analyzed (Participants) | 0 | 1
  Subject 6 (week 6) |  | 0.12
  Subject 7 (week 5): number analyzed (Participants) | 0 | 1
  Subject 7 (week 5) |  | 0.44
  Subject 7 (week 6): number analyzed (Participants) | 0 | 1
  Subject 7 (week 6) |  | 1.27
  Subject 8 (week 5): number analyzed (Participants) | 0 | 1
  Subject 8 (week 5) |  | 0.00
  Subject 8 (week 6): number analyzed (Participants) | 0 | 1
  Subject 8 (week 6) |  | 0.29
  Subject 10 (week 5): number analyzed (Participants) | 0 | 0
  Subject 10 (week 6): number analyzed (Participants) | 0 | 0
  Subject 12 (week 5): number analyzed (Participants) | 0 | 0
  Subject 12 (week 6): number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to final study date per patient, approximately 10 months.
Arm/Group | Non Surgical-Radiation Only | Malignant Tumor Surgery And Radiation
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/10
Other Adverse Events (participants affected / at risk) | 0/2 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Surgical-Radiation Only (N=2) | Malignant Tumor Surgery And Radiation (N=10)
Allergic reaction (General disorders) | 0 (0) | 1 (1) — Patient had an allergic reaction to then non-investigational FDA approved bone labeling drugs (demeclocycline).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02323295/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02323295/ICF_001.pdf